CLINICAL TRIAL: NCT01006109
Title: Recording and Modulation of Neuronal Mechanisms During Operant Conditioning: A MEG Study
Status: Terminated | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 100003; 10-N-0003
Record Dates: First submitted 2009-10-30; First posted 2009-11-02 (Estimated); Last update posted 2019-12-17 (Actual); Status verified 2017-09-07

CONDITIONS: Central Nervous System
Keywords: MEG; Repetitive TMS (rTMS); Decision-Making; Healthy Volunteers; HV; Healthy Volunteer

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional

SUMMARY:
Background:

- Most of the time, humans make decisions according to their consequences, especially if they will be beneficial, and will avoid or try to avoid doing an action if it has a bad outcome. The way that the brain prepares a movement has been studied in detail, but the way the brain makes decisions before carrying out an action is still poorly understood. Researchers are interested in learning more about the decision-making process and how it affects the brain.

Objectives:

- To record the activity of the brain during decision-making processes.

Eligibility:

- Healthy, right-handed volunteers between 18 and 40 years of age.

Design:

* Potential participants will have a screening visit with a medical history and neurological examination to determine eligibility.
* This study requires seven visits: one magnetic resonance imaging (MRI) visit and 6 magnetoencephalography (MEG) recording visits. The MEG recording visits will include transcranial magnetic stimulation (TMS). All visits will be spaced at least 1 week apart. Total participation will last about 6 weeks.
* Participants will have an MRI scan at the first study visit.
* The MEG procedures will record brain activity during a series of computer tests involving winning or losing money. TMS will be performed during these visits, separate from the test....

DETAILED DESCRIPTION:
Objective:

The objective is to study cerebral activity associated with reward-related decision making. We plan to analyze and localize electrical activity of the brain related to such processes with magnetoencephalography (MEG). We also want to modulate the activity of these areas using repetitive transcranial magnetic stimulation (rTMS). We would like to analyze the consequences of these procedures on both brain activity and behavioral performance. This protocol will provide new information on cortical regions involved in decision-making and how these areas communicate with one another.

Study population:

50 right-handed adult healthy volunteers.

Design:

A probabilistic reversal task will be performed: subjects will have to choose between pairs of stimuli associated with changing probabilities of rewards and losses. Using MEG, their cerebral activity will be recorded during task performance.

Since we want to modulate the cortical activity of cerebral areas involved in reward-related decision making, the study will be carried out in 8 different visits (screening visit, structural MRI acquisition and 6 recordings visits). In one visit, decision-making will be studied with no previous cortical stimulation. In 3 visits, decision-making will be studied after stimulation of one of 3 regions of interest. In one visit, decision-making will be studied after stimulation of a cortical area that is not thought to be involved in the process. Lastly, decision-making will be analyzed following a sham stimulation to test a possible placebo effect of rTMS.

Outcome measures:

Outcome measures are as follow:

1. Task-related: reaction time and error rate during the task performance.
2. MEG signal: scalp and source coherence between cortical regions, amplitude and latency of event-related potentials and even-related (de)synchronization.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Aged 18 to 40 years
  2. Right-handed (Edinburgh Handedness Quotient greater than 60).

EXCLUSION CRITERIA:

1. Abnormal neurological exam, current or past history of neurological disease or psychiatric disease. Patients with neurological diseases of the central nervous system that impair the motor system or cognitive function will be excluded. Patients with axis I psychiatric disorders will be excluded. Such disorders will be identified or suspected on neurologic examination. If there is any uncertainty about a possible psychiatric diagnosis, psychiatric consultation will be obtained.
2. Use of antidepressants, anxiolytics, anticonvulsants, antipsychotics, antiparkinson drugs or stimulants during the 3 months prior to their screening visit, and/or hypnotics or antihistamines during the 1 month prior to their screening visit
3. Having a pacemaker, an implanted medical pump, a metal plate or metal object in the skull or eye (for example, after brain surgery), or a history of seizure disorder
4. Pregnancy
5. Any contraindication to scanning on the NMR Center MRI safety screening questionnaire: cardiac pacemaker; implanted cardiac defibrillator; aneurysm clip; neuro or bone stimulator; insulin or infusion pump; implanted drug infusion device; cochlear, otologic, or ear implant; prostate radiation seeds; IUD (intrauterine device); transdermal medication patch (Nitro); any type of prosthesis (eye, penile); heart valve prosthesis; shunt (spinal/intraventricular); wire sutures or surgical staples; bone/joint pin, screw, nail, plate; body tattoos or makeup (eyeliner/lip); body piercing(s) (non-removable); breast tissue expander; any metallic implants or objects.
6. Metallic dental fillings that are likely to cause MRI artifacts
7. Claustrophobia
8. Inability to give informed consent
9. Personal or family history of hearing loss

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2009-10-22; Study Completion 2017-09-07

PRIMARY OUTCOMES:
Performance of each subject, before and after each cTBS session. We will measure their reaction time and the number of errors which corresponds to the number of times the subject did not choose the target which could have made him/her win money... | During the MEG recording

SECONDARY OUTCOMES:
MEG signal: latency and amplitude of evoked and induced activity related to decision-making, without and after cTBS. The cerebral sources of these activities will also be computed and their interaction will be studied using source coherence ana... | During the MEG recording

CONTACTS AND LOCATIONS:
Overall Officials: Mark Hallett, M.D., Principal Investigator — National Institute of Neurological Disorders and Stroke (NINDS)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Andrew C, Pfurtscheller G. Event-related coherence as a tool for studying dynamic interaction of brain regions. Electroencephalogr Clin Neurophysiol. 1996 Feb;98(2):144-8. doi: 10.1016/0013-4694(95)00228-6. PMID 8598174
- [Background] Andrew C, Pfurtscheller G. Dependence of coherence measurements on EEG derivation type. Med Biol Eng Comput. 1996 May;34(3):232-8. doi: 10.1007/BF02520079. PMID 8762831
- [Background] Brandt SA, Ploner CJ, Meyer BU, Leistner S, Villringer A. Effects of repetitive transcranial magnetic stimulation over dorsolateral prefrontal and posterior parietal cortex on memory-guided saccades. Exp Brain Res. 1998 Jan;118(2):197-204. doi: 10.1007/s002210050272. PMID 9547088